CLINICAL TRIAL: NCT03324724
Title: Integrative Cognitive-Affective Therapy for Adolescent Eating Disorders (ICAT-A)
Brief Title: Integrative Cognitive-Affective Therapy for Adolescent Eating Disorders
Acronym: ICAT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Eating Disorders Association (Other)
Responsible Party: Principal Investigator, Jocelyn R. Lebow, Ph.D., L.P., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-008708
Record Dates: First submitted 2017-09-05; First posted 2017-10-30 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Eating Disorder; Emotional Disorder
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with Eating Disorder (Experimental): Adolescents with bulimia nervosa or binge eating disorder, with one or more of their parents, will receive integrative cognitive-affective therapy for adolescents (ICAT-A).
  Interventions: Behavioral: Integrative cognitive-affective therapy for adolescents (ICAT-A)

INTERVENTIONS:
Behavioral: Integrative cognitive-affective therapy for adolescents (ICAT-A) — Participants will receive a 21-session individual psychotherapy approach with 4 phases. In addition, there will be 7-13 additional conjoint parent sessions.

SUMMARY:
Recently, Integrative Cognitive-Affective Therapy (ICAT), a novel intervention for bulimia nervosa (BN) and binge eating disorder (BED) that targets emotion regulation deficits, has shown promise in reducing eating disorder symptoms as well as improving emotion regulation capacities in adults. However, this treatment has not been investigated in an adolescent sample. Given the contributing role of emotion regulation in adolescent eating disorder symptoms and limited treatment options for adolescents with BN and BED, the aim of this study is to adapt the existing adult ICAT treatment for adolescents with clinically significant binge eating (ICAT-A) and to evaluate the extent to which ICAT-A is helpful in reducing binge eating and associated eating disorder symptoms in a younger sample.

ELIGIBILITY:
Inclusion Criteria:

* Subject with full and sub-threshold bulimia nervosa and binge eating disorder (that is binge eating weekly)
* No major weight loss (defined as a reduction of 10% baseline body weight or more)
* Subject who meet criteria for any Diagnostic and Statistical Manual of Mental Disorders (DSM-5) eating disorder characterized by binge eating with or without compensatory behavior
* Subjects who take medications that do not directly impact weight or appetite (including Selective serotonin reuptake inhibitors (SSRI) antidepressants) will be included if their dose has been stable for at least six weeks
* Subject must be living at home
* At least one parent/guardian is willing to participate in the treatment.

Exclusion Criteria:

* Subject on medications that influence weight or appetite (including antipsychotic medications)
* Subject who is medically or psychiatrically unstable (defined as requiring hospitalization within the past 3 months)
* Acutely suicidal requiring current hospitalization or who meet criteria for substance use disorder in the past month
* Subjects who become or psychiatrically unstable during the study will be re-evaluated, removed from the study, and referred for appropriate treatment.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Change in Eating Disorder Examination (EDE) | baseline, end of treatment (approximately 8 months)
  The EDE is a semi-structured interview conducted by a trained clinician to assess the psychopathology associated with the diagnosis of an eating disorder. The EDE is rated through the use of four subscales and a global score. The four subscales are: 1) Restraint, 2) Eating concern, 3) Shape concern, 4) Weight concern. The questions concern the frequency in which the patient engages in behaviors indicative of an eating disorder over a 28-day period, but some questions extend out to cover the previous 3 months. To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscale. To obtain an overall score, the four subscales scores are summed and the resulting total divided by the number of subscales (4). The total score can range from 0 (normal) to 6 (high eating disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn R Lebow, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials